CLINICAL TRIAL: NCT01452126
Title: Minimum Effective Anesthetic Concentration of Supraclavicular Block, Infraclavicular Block, Femoral Nerve Block and Sciatic Nerve Block Via the Popliteal and Parasacral Approach
Brief Title: Minimum Effective Concentration of Ropivacaine for Brachial Plexus Block Via the Supraclavicular and Infraclavicular Approach, Femoral Nerve Block, Sciatic Nerve Block Via the Popliteal and Parasacral Approach
Acronym: MEAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Departure of principal investigator
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Timothy R Petersen, Research Information Specialist, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: UNM HRRC 11-030
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Surgical Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ropivacaine (Experimental): Sequential allocation of ropivacaine concentration depending on the success or failure of surgical anesthesia of the previous patient
  Interventions: Drug: Ropivacaine concentration

INTERVENTIONS:
Drug: Ropivacaine concentration — Single shot preoperative perineural injection of ropivacaine to achieve surgical anesthesia. The concentration of ropivacaine is lowered by 0.05% after every successful surgical anesthesia specific to that block and raised by 0.05% after every unsuccessful surgical anesthesia specific to that block

SUMMARY:
This is a dose finding study to identify the minimum effective anesthetic concentration (MEAC) of ropivacaine to produce insensate body parts sufficient for surgery in supraclavicular and infraclavicular approaches to the brachial plexus, parasacral and popliteal approaches to the sciatic nerve, femoral nerve and transversus abdominis plane (TAP) blocks in adults.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I to III (patients may be healthy or have systemic disease, but any disease does not pose a constant threat to life, and patients are neither moribund, nor not expected to survive without the operation).
* Age 18 or above
* Undergoing elective ambulatory surgery of the upper limb (excluding the shoulder), lower limb (excluding the hip), or lower abdomen with sensory blockade as part of the pain management plan.

Exclusion Criteria:

* Body mass index of >35 kg/m2 (higher chance of failure)
* Deformities of the leg (for patients in the parasacral, femoral, and popliteal groups), or the chest or shoulder (for patients in the supraclavicular, infraclavicular, and TAP groups)
* Preexisting infection at the injection site
* Existing neurologic disease
* Allergy to local anesthetic agents
* Severe respiratory disease
* Coagulopathy
* Any other contraindication to the block being considered
* Patients requiring total motor blockade as well as sensory blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, MD, Principal Investigator — University of New Mexico
Locations (1):
- Univeristy of Mexico Outpatient Surgical and imaging service, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ropivacaine: Each patient received ropivacaine-based nerve blockade at a fixed volume, with concentration determined per protocol
Arm/Group | Ropivacaine
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 19
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Effective Concentration of Ropivacaine to Produce Surgical Anesthesia in 50% of Population
Description: The concentration of ropivacaine for each patient's nerve-block injection was determined per protocol.
Time Frame: 1 day
Measure: Number; unit: percentage concentration, ropivacaine
Groups:
- Femoral Nerve Block: Ropivacaine-based blockade of the femoral nerve, with concentration per protocol.
- Supraclavicular Blockade: Ropivacaine-based blockade of the brachial plexus nerves via a supraclavicular approach, with concentration per protocol.
- Infraclavicular Blockade: Ropivacaine-based blockade of the brachial plexus nerves via an infraclavicular approach, with concentration per protocol.
- Popliteal Nerve Block: Ropivacaine-based blockade of the popliteal nerve, with concentration per protocol.
Arm/Group | Femoral Nerve Block | Supraclavicular Blockade | Infraclavicular Blockade | Popliteal Nerve Block
Number analyzed (Participants) | 14 | 13 | 11 | 11
percentage concentration, ropivacaine | 0.09 | 0.11 | 0.16 | 0.37

2. Secondary Outcome: Number of Patients With Complications
Description: All patients were followed up for complications such as bleeding, infection, side effects, nerve damage
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine
Number analyzed (Participants) | 49
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Ropivacaine
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 11/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine (N=49)
Failure of regional anesthesia (Surgical and medical procedures) | 11 (11) — As this was a dose-finding study, it was expected that some patients would experience failure of regional anesthesia.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Confidence intervals for primary outcome are not reliable and therefore not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes